CLINICAL TRIAL: NCT00699595
Title: Hormonal Effects on Pain Perception
Acronym: HEPP
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Froelich, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F070721003
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy; Progesterone Levels; Pregnancy Associated Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Plasma for progesterone levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Term pregnant women: Healthy women scheduled for elective Cesarean section.

SUMMARY:
To investigate if labor pain is affected by mother's hormone levels.

The hormonal effects of pregnancy are well documented. Although differences in pain sensitivity between women and men are partly attributable to social conditioning and to psychosocial factors, many laboratory studies of humans have described sex differences in sensitivity to noxious stimuli, suggesting that biological mechanisms underlie such differences. Some animal studies have suggested that sensitivity to pain decreases during pregnancy because of the progressive activation of endogenous pain inhibitory systems. This effect may be mediated by pregnancy-associated hormones, in particular progesterone.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women at term (>37GA)

Exclusion Criteria:

* chronic pain
* regular analgesic medication
* severe cardiopulmonary problems
* very difficult intravenous access
* advanced labor
* precipitous delivery

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy term pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in heat pain threshold and tolerance | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael Froelich, MD, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States